CLINICAL TRIAL: NCT02447731
Title: The Effects of Sound Energy on Pulmonary Gas Exchange
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator passed away.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: Sound Energy
Record Dates: First submitted 2015-02-02; First posted 2015-05-19 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure
Keywords: respiratory insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sonic Gas Exchange: Gas exchange rates in the lungs of subjects breathing through a mouthpiece will be compared with their gas exchange rates after addition of sound pressure vibrations into the supplied gas. 'Induction of sound waves in lungs by "sonic oscillator"' can be as loud as a human screaming or singing very loudly (about 95 dB). The effects of these pressure oscillations on gas exchange will be assessed using 3 tests as explained in the section under "detailed description".
  Interventions: Device: Induction of sound waves in lungs by "sonic oscillator"

INTERVENTIONS:
Device: Induction of sound waves in lungs by "sonic oscillator" — A device called sonic oscillator will add sonic waves to the inhaled gases while the subjects are going through 3 tests measuring the variations made in pulmonary functions induced by sound waves.
  Other Names: Sonic Lung Ventilation

SUMMARY:
Study of the effects of sonic pressure oscillations on pulmonary gas exchange with added dead space.

DETAILED DESCRIPTION:
Sound waves are used in various industries to accelerate the process of mixing or separating fluids (gases/liquids). We have proved that certain sound waves can safely improve gas exchange in the lung of rats through accelerating gas diffusion inside their airways and alveoli. Now we want to see if similar sound waves can improve gas exchange in humans.

The device which creates the sound waves is a sonic pressure oscillator capable of making sound waves similar in loudness and frequency to loud human singing or screaming. These waves are mainly in the frequency range of 50-500 Hz (Hertz, oscillations per second) with intensity of 85-105 dBs (deci Bells, unit of sound pressure intensity).

We performed two bench top studies and witnessed the ability of sound waves to augment gas diffusion. In a pilot study in rats we showed a safe and significant improvement in pulmonary gas exchange under influence of sound energy. The effects of sound waves on gas exchange in a human subject, the principle investigator (PI), was also analyzed in a metabolic test with promising results. A clinically significant improvement in the PI's pulmonary gas diffusion was also noted in a DLCO (diffusing lung capacity for carbon monoxide) test. On yet another test, artificially enlarged pulmonary dead space study, the PI's transcutaneous oxygen and carbon dioxide pressures (PtcCO2 & PtcO2) were measured and results were indicative of presence of desired and safe effects of particular sound waves in pulmonary gas exchange. The above mentioned studies support the rationale, objectives, and methodology of the proposed studies.

Our human studies will be composed of a primary and a secondary part. In the primary part, the sound waves are not introduced into the subjects' lungs directly and they are rather delivered into an open end cylinder while the subjects breathe the air from the closed end of the cylinder. The sound intensity will be kept in the range of 95-105dB.

In the second part of the studies, the sound waves of lower intensity (85-95dB) are directly introduced into the subjects' lungs while the subjects are going through 1) a metabolic test and 2) a lung diffusion capacity (DLCO) test. The results of these tests will be compared to the subject's baseline test results (without sound waves).

In both parts of the study, the subjects' nostrils will be clamped by ordinary plastic nose clamps as they will be asked to hold a mouthpiece and breathe through it.

In the primary part, sound waves of 95-105dB will be delivered into a 16 L (liter) frustum (conical cylinder). The frustum's wider base is open to room air but its smaller base is closed. A 2x20 cm tube will connect the closed end of the frustum to the mouthpiece. The subjects will be breathing in and out of the narrower (closed) base of the frustum through the mouthpiece for 3 minute cycles followed by 3 minute cycles of breathing fresh room air. The subjects' PtcCO2 and PtcO2 will be measured with the frustum held in various spatial orientations in regard to its open base which will be 1) vertical upward (+90 degrees with horizon), 2) horizontal (0 degrees), vertical downward (-90 degrees), and tilted to -45 degree angles. This test will take at least 6x4=24 minutes, and not more than 30 minutes for each subject. Then same tests will be done with sound energy introduced into the frustum. Total time for studying each subject will be approximately 48-60 minutes.

Secondary part of the study is composed of two sections. In the first section, diffusion capacity of the lungs will be measure while the sound waves are being played by the transducer and delivered via a mouth piece into the subjects' oral cavity. The sound waves will be travelling down the pulmonary airways and into the alveoli. An examiner will listen to the chest wall to make sure that the subject is allowing the waves to travel down the airways without obstructing the path to the sound waves by inadvertently holding the tongue up or holding breath. Said mouth piece is connected via a Y-connector to the DLCO machine and the tube which delivers the sound waves. The duration of exerted sound effect will be only 9 seconds as per protocol of a routine DLCO testing. This period coincides with the time when the subject is taking a deep breath and holding it for 9 seconds. Lung diffusion capacity of the subjects will be measured and compared with soundless test results. Although the test uses very small amount of carbon monoxide (CO) as the tracer gas but the amount is considered negligible and quite safe. This test has been done in humans routinely for many years with no known discernible side effects. It has been approved by FDA many years ago. There is an abundance of medical literature regarding the safety and methods used in DLCO. There are also multiple YouTube videos showing how DLCO is done. We will encourage the participants to watch these videos before the studies. The subjects will be sitting comfortably on a chair and holding the mouth piece in their mouths and breathing the room air. They can easily interrupt the test at any time by simply taking the mouthpiece out of their mouths.

In the second section, subjects will go under metabolic tests where their exhaled oxygen (O2) and carbon dioxide (CO2) are measured with and without sound effects. Metabolic tests have been approved by FDA for many years and are generally considered very safe. During the test, the participants breathe from the mouth piece with their nostrils clamped. Breathing gases will be provided by connecting the mouth piece to a tube which usually has a base flow of room air 40L/min or more. In order to show oxygenation improvement via sound energy we will have to create a suboptimal respiratory environment and artificially induced hypoxia. Mild hypoxia is generally well tolerated by healthy humans although it might make the individual feel short of breath and tachypneic. We will add nitrogen to the supplied air to bring the fraction of inhaled oxygen (FiO2) down to 17.5% which correlates breathing at an altitude of 7500 feet (approximately 2250m), or similar to a ski resort, except that we don't ask our subjects to get involved in vigorous exercise like skiing, and the test is only ~20 minutes. The lowered FiO2 will bring the subjects' pulse ox (SpO2) down to 92-94% which is generally considered safe and well tolerated by all normal human subjects with no cardiopulmonary conditions. The resultant mild and transient respiratory alkalosis has no clinical significance as it only involves a 20 minute test and the pH imbalance would be buffered naturally without inducing any electrolyte abnormalities.

The acoustic transducer, as mentioned briefly earlier, is a simple sound wave generator and is composed of a tone generator (usually a computer), an electronic amplifier, an acoustic transducer similar to an ordinary loudspeaker, and a funnel and tubing system that directs the sound waves into the subjects' mouthpiece. Its function is very similar to standing in front of a loudspeaker and letting the sounds penetrate into the mouth/nose and down the pulmonary airways except that in order to protect the ears and intensify the sounds a funnel is used to capture the waves and direct them into the oral cavity via a tube. The device is made, tuned, and calibrated by the principal investigator. It can produce tones from 20 Hz to about 11 KHz with useful intensities ranging from 65dB to a maximum of 110dB. The simple device has been successfully used in rats and a human (PI) without any discernible side effects.

For more detailed description of the methodology and results of our previous studies please refer to the attached documents with the referenced literature.

Data Collection:

During the first part of the study, data with subjects' PtcCO2, PtcO2, heart rate, respiratory rate, minute volume, and blood pressure will be logged onto a spread sheet and saved on password protected computers.

Lung diffusion capacity variations under the influence of sound vibrations will be measured and recorded using a DLCO machine at the respiratory department of LLUMC. Data will also be saved on password protected computers using encrypted MS-Excel in addition to the memory of the DLCO machine. During the metabolic tests, inhaled and exhaled concentrations of O2 and CO2 will be continuously monitored along with subjects' heart rate, breath rate, pulse oxymetry, blood pressure, general comfort level of the subject and his/her clinical well being. The encrypted and password protected data will be collected on Microsoft Spreadsheets for statistical analysis by a biostatistician.

RISK AND INJURY:

Human ears are particularly prone to damage by loud sounds. Ear pain or discomfort can happen at sound levels as low as 110dB but painful sound levels are generally considered to be in the range of 125-135dB. Other organs tolerate sound wave much better and tissue damage normally does not occur in sound intensity levels less than 160-170dB. Sound intensity will be monitored and recorded during the studies. The intensities will always be kept to below 105dB which is significantly below any harmful levels considering the fact that sound pressure levels are measure in logarithmic scale.

During the metabolic tests, the subjects pulse oximetry will be kept above 92% to avoid any ill effects. These levels are very well tolerated by humans and ordinarily physicians do not supplement any oxygen to patients at these levels. Very brief hypoxia with hypercapnia will happen during the frustum test when the frustum is held at held at +90 degree position as the SpO2 will plummet to upper 70s to lower 90s in about 3 minutes which is the limit of this test. We will halt the test before the 3 min landmark if a subject's SpO2 went below 80%. The brief and transient hypoxia and hypercapnia is well tolerated. A medical doctor will be present at all times whenever the tests are running. A thorough medical exam immediately before the tests will secure safety of the subjects as well.

Metabolic studies and DLCO tests have been done routinely for many years/decades and are generally considered very safe. The amount of inhaled carbon monoxide used as a tracer gas in DLCO is significantly below any toxic levels. These tests have been approved by FDA for a long time and are considered safe even in patients with pulmonary disorders.

BENEFITS:

The studies do not have any direct or immediate benefit to the subjects participating in the study. It has been anticipated that sound waves may help decrease incidence and severity of "ventilation induced lung injury or VILI" to an extent yet to be measured. The main reason behind this postulation is that addition of proper sound waves to breathing gases will enable us to effectively ventilate lungs with lower FiO2 and/or less mean airway pressure (Pmaw) compared to the currently available technologies. It is known for a long time that high FiO2/Pmaw are the two major predictors of VILI. It is also anticipated that the outcome of cardiopulmonary resuscitation (CPR) and many acute or chronic pulmonary disorders such as COPD, asthma, cystic fibrosis, bronchopulmonary dysplasia, restrictive lung disorders, acute lung injury, pneumothorax, RDS, and some other conditions may improve through use of proper sound waves.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers in the age group.

Exclusion Criteria:

* Any acute or chronic cardiopulmonary disorder including a simple common cold.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy adults of any gender.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Percent Improvement in PtcO2 & PtcCO2 | 1 month
  Sonic vibrations similar to human screaming should improve pulmonary gas diffusion by more than 5% in few seconds.

SECONDARY OUTCOMES:
mL/min exhaled VCO2 and VO2 | 1 month
  VO2 and VCO2 in exhaled gas will be measured in mL/min to see if the values increase with sound energy introduced into the lungs intermittently with 2 minutes sound on and 2 minute sound off. Any increase will show how much improvement in oxygen uptake and carbon dioxide liberation is achieved with sound vibrations similar to human loud singing or screaming.

OTHER OUTCOMES:
Percent improvement in lung diffusion capacity | 1 month
  lowest tolerable fraction of inhaled oxygen under influence of sound energy will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M. R. Jam, MD, Principal Investigator — Assistant Professor
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States